CLINICAL TRIAL: NCT00654459
Title: Effects of Armolipid Plus on Cholesterol Levels and Endothelial Function
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Collaborators: Rottapharm (Industry)
Responsible Party: Serafino Fazio MD, Federico II University
Other Study IDs: ARM 02-07
Record Dates: First submitted 2008-04-02; First posted 2008-04-08 (Estimated); Last update posted 2008-04-16 (Estimated); Status verified 2008-04

CONDITIONS: Hyperlipidemia; Endothelial Dysfunction
MeSH Terms: conditions — Hyperlipidemias | interventions — policosanol

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- A
  Interventions: Dietary Supplement: Mixture of Berberine, Policosanol, Red Yeast, Placebo
- B
  Interventions: Dietary Supplement: Mixture of Berberine, Policosanol, Red Yeast, Placebo

INTERVENTIONS:
Dietary Supplement: Mixture of Berberine, Policosanol, Red Yeast, Placebo — A tablet one a day for 6 weeks
  Other Names: Armolipid Plus

SUMMARY:
Some nutraceuticals are often advised for their lipid lowering effects. Although many clinical trials have been conducted to assess their efficacy many doubts remain whether they could be considered an effective alternative to statins therapy.

The aim of this study was to evaluate the lipid lowering effects and the improvement of endothelial dysfunction in patients with hyperlipidemia, treated with a nutraceutical product (Armolipid Plus)

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged between 18 and 70
* Total cholesterol levels > 220 mg/dl and LDL-Cholesterol > 130 mg/dl;
* Patients with concomitant pathology such as diabetes, chronic heart failure, coronary artery disease, arterial hypertension, dysthyroidism, were admitted as long as stable in the previous three months

Exclusion Criteria:

* Proven intolerance to an Armolipid Plus compound
* Pregnant women, and women planning to conceive
* Patients in therapy with lipid lowering drugs within the previous 6 weeks
* Triglycerides concentration > 500mg/dl were excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: males and females aged between 18 and 70 with hypercholesterolemya
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2007-07; Primary Completion 2008-01 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure of this study was the percentage change from baseline of total cholesterol (C), LDL- cholesterol (LDL-C), HDL-cholesterol (HDL-C),and Triglycerides (Tg) plasma concentrations. | 6 weeks

SECONDARY OUTCOMES:
Secondary end point included improvement of endothelial dysfunction assessed by an echo flow mediated distribution test. | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Serafino Fazio, MD, Principal Investigator — Federico II University
Locations (1):
- Department of internal medicine University Federico II, Naples, Italy